CLINICAL TRIAL: NCT02747303
Title: The Clinical Relevance of Margins in Frameless Stereotactic Radiosurgery for Intact Brain Metastases: a Randomized Trial of 0 vs 2 mm Margins
Brief Title: Frameless Stereotactic Radiosurgery for Intact Brain Metastases
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB15-1476
Record Dates: First submitted 2016-04-19; First posted 2016-04-21 (Estimated); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Brain Metastases
Keywords: brain metastases; Stereotactic Radiosurgery
MeSH Terms: conditions — Brain Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stereotactic Radiosurgery to 2 mm GTV to PTV margins (Active Comparator)
  Interventions: Procedure: Stereotactic Radiosurgery
- Stereotactic Radiosurgery to 0 mm GTV to PTV margins (Experimental)
  Interventions: Procedure: Stereotactic Radiosurgery

INTERVENTIONS:
Procedure: Stereotactic Radiosurgery — The SRS dose will depend on the maximum diameter of the gross tumor volume (GTV)

SUMMARY:
This is a randomized study to determine if not treating planning target volume (PTV) margins during radiation therapy worsens progression free survival rates in patients with brain metastases.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 18 years old) with an ECOG Performance Status 0-2 and a life expectancy of 3 months or more.
* Histologically confirmed systemic malignancy with gadolinium contrast-enhanced MRI scan demonstrating 1-5 intraparenchymal brain metastases.
* Well-circumscribed, measureable intraparenchymal brain lesion(s) with maximum tumor diameter ≤3.0 cm. If multiple lesions are present, the other(s) must not exceed 3.0 cm in maximum diameter. At least one lesion must be ≥1.0 cm in maximum diameter and ≥0.5 cm in a perpendicular diameter to be considered measurable disease.
* Negative urine or serum pregnancy test done ≤ 14 days prior to CT simulation, for women of child-bearing potential only.
* Ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria:

* Diagnosis of germ cell tumor, small cell carcinoma or hematologic malignancy.
* Metastases in the brain stem, midbrain, pons, medulla, or within 7 mm of the optic apparatus (optic nerves, chiasm and optic tracts).
* Diagnosis of leptomeningeal disease.
* Prior cranial radiotherapy within 90 days of trial enrollment or prior SRS at any time to any lesion to be treated on protocol
* Chemotherapy (including oral agents and targeted agents) or immunotherapy given within 14 days of SRS. Hormonal therapy is permitted. For Her2+ breast cancer patients, anti-Her2 therapy cannot be given within 14 days of SRS. Patients who are scheduled to receive trastuzumab emtansine after SRS cannot be enrolled.
* Contraindications to gadolinium contrast-enhanced MRI (eg, non-compatible pacemaker, eGFR<30, gadolinium allergy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Estimated)
Dates: Start 2023-09-05 (Actual); Primary Completion 2028-08-22 (Estimated); Study Completion 2028-08-22 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) rates estimated by the Kaplan-Meier method at 6 months | 6 months
  Progression free survival (PFS) rates will be estimated by the Kaplan-Meier method and the 0-mm and 2-mm groups will be compared via the log-rank statistic with a one-sided test of significance, using follow-up data up to 6 months.

SECONDARY OUTCOMES:
Progression free survival (PFS) rates estimated by the Kaplan-Meier method | 2 years
  Progression free survival (PFS) rates will be estimated by the Kaplan-Meier method and the 0-mm, and 2-mm groups will be compared via the log-rank statistic with a one-sided test of significance, using follow-up data up to 6 months.
Overall survival rates | 2 years
  Time from Stereotactic Radiosurgery (SRS) completion to death.
Rates of radiation necrosis | 2 years
  To evaluate the superiority of frameless LINAC-based SRS using 0 mm margins compared to 2 mm margins in reducing rates of radiation necrosis.
Rates of pseudoprogression | 2 years
  To evaluate the superiority of frameless LINAC-based SRS using 0 mm margins compared to 2 mm margins in reducing rates of radiation pseudoprogression.
Local failure rates | 2 years
  Local failure and OS rates at 6 months, 1 year and 2 years will be estimated by the Kaplan-Meier method, comparing arms via the log-rank statistic.
Rate of acute central nervous system (CNS) Common Terminology Criteria for Adverse Events (CTCAE) v4.0 grade 2 and higher toxicities | 90 days
  Any acute CTCAE v4.0 CNS Grade 2+ and Grade 3+ toxicities, within 90 days of SRS completion (toxicity must be specified).
Rate of late central nervous system (CNS) Common Terminology Criteria for Adverse Events (CTCAE) v4.0 grade 2 and higher toxicities | 2 years
  To compare rates of late (greater than 90 days from SRS) CTCAE v4.0 CNS Grade 2+ and Grade 3+ toxicities.
Rates of distant intracranial failure | 2 years
  The appearance of new non-target lesions ≥5 mm following completion of radiotherapy will be considered distant intracranial failure. If a non-target lesion <5 mm is found on a later scan to have increased to ≥ 5 mm, distant intracranial failure will be declared at the date of the earliest scan showing the new lesion.
Rates of salvage therapy | 2 years
  Time to initiation of any combination of salvage Stereotactic Radiosurgery (SRS), Whole Brain Radiation Therapy WBRT, or neurosurgical resection for intracranial failure.
Association between dose and risk of radionecrosis or pseudoprogression | 2 years
  To determine association between V10Gy and V12Gy all tissue, whole brain and normal brain parameters and risk of radionecrosis or pseudoprogression.

CONTACTS AND LOCATIONS:
Overall Officials: Steven J. Chmura, M.D., Ph.D., Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States